CLINICAL TRIAL: NCT02309710
Title: Prospective Study of Male Circumcision Using the ShangRing Device in Routine Clinical Settings in Malawi
Brief Title: Male Circumcision (MC) Using the ShangRing™ Device in Malawi
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 595330-3
Record Dates: First submitted 2014-11-21; First posted 2014-12-05 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Male Circumcision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ShangRing (Experimental): ShangRing administered to men seeking medical male circumcision
  Interventions: Device: ShangRing

INTERVENTIONS:
Device: ShangRing — ShangRing administered to males seeking medical male circumcision

SUMMARY:
This prospective study will evaluate the safety and acceptability of the ShangRing device for medical male circumcision (MMC) during routine service delivery in Namitete, Malawi

DETAILED DESCRIPTION:
Although voluntary medical male circumcision (VMMC) was adopted as a prevention strategy in 2011, MMC prevalence in Malawi is low with estimates between 2 and 20%. The 5-year national VMMC target for Malawi is 80% of men ages 15 - 49, or more than two million procedures. Since 2011, only 42,700 VMMCs have been done for HIV prevention, about 2% of the target. Of the 29 healthcare districts in Malawi, only a minority are supported by non-governmental (NGO) and U.S. government-funded VMMC programs. Major obstacles include few VMMC service-delivery points; few trained service providers; poor availability of prepackaged disposable VMMC kits requiring re-use of instruments and supplies; few organized campaigns or community mobilization programs; and drop-in services only.

Scale-up of adult MMC services in Malawi could be accelerated by the availability of simplified, bloodless methods. Methods of MMC using devices may also increase safety, efficiency and acceptability. Although many devices are available and widely used for infant circumcision, fewer devices exist for use in adult male circumcision and there are limited data on device use in adults. Small-scale safety studies, randomized controlled trials (RCTs), and field demonstration studies are required before the safety, effectiveness, acceptability, and feasibility of any device is assured.

Several devices have recently been developed that have the potential to simplify and shorten both training time and surgical duration by eliminating the need for suturing and hemostasis as well as allow for task-shifting to lower-level cadres of healthcare providers (i.e. non-physician), thereby reducing the strain on healthcare systems by having more healthcare workers available to provide MMC services. One such device is the ShangRing.

In the WHO framework, smaller bridging studies are recommended to address additional questions about particular sub-populations and specific conditions of use (WHO 2011). This research study will assess the safety and acceptability of the ShangRing within the context of routine service delivery in Namitete, Malawi. The investigators will enroll 500 HIV-uninfected adult men aged 18 to 49 years voluntarily seeking medical male circumcision. The men will be scheduled for two follow-up visits at 7 and 42 days after ShangRing placement for device removal and a healing check, respectively. Results from this study will inform the Malawi Ministry of Health (MOH) as it decides on the integration of MMC devices into its national VMMC program.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 18 to 49 years;
* Must be HIV-uninfected per same-day routine HIV testing and counseling (HTC) at the clinic;
* Must be uncircumcised (on examination);
* Must be in good general health, at the discretion of the clinician;
* Must be free of genital ulcerations or other visible signs of sexually transmitted infections(STI) on examination;
* Must be able to understand study procedures, and agree to abide by them including the follow-up visit schedule;
* Must be able to communicate in English or Chichewa;
* Must freely consent to participate in the study, be available for follow-up visits, and sign a written informed consent form (ICF); and
* Must provide full contact information including cell phone number, address, and other locator information

Exclusion Criteria:

* Has an anatomic abnormality (e.g. phimosis or hypospadias) that contraindicates ShangRing MMC;
* Takes a medication that would be a contraindication for elective surgery, such as an anticoagulant or steroid;
* Has a self-reported medical condition that would be a contraindication for elective surgery, e.g. hemophilia, extreme obesity, poorly controlled diabetes, sickle cell anemia;
* Has a self-reported allergy or sensitivity to lidocaine or other local anesthesia; or
* Is not available to be circumcised on the same day as screening.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The percentage of men with moderate and severe adverse events will be tabulated with 95% confidence intervals | up to 42 days following circumcision procedure

SECONDARY OUTCOMES:
proportion of men ineligible for MMC with ShangRing | up to four months
  The proportion and 95% confidence interval (CI) of men who did not receive ShangRing circumcision because of inability to find an appropriate size will be reported
Percentage distribution of overall satisfaction for study participants | at Day 42 visit
  Study participants will be interviewed using a standardized questionnaire with items on overall satisfaction with the ShangRing procedure.
Percentage preference for ShangRing procedure among study MC providers | an expected average of one month after study initiation
  Study circumcision providers will complete the first questionnaire after receiving training and completing 20 circumcision and device removal procedures. Providers will be interviewed using a standardized questionnaire that includes items on preference for ShangRing.
Complete Healing at final follow up visit | up to 42 days
  Percentage of men with complete healing at 42 days for all study participants
Percentage preference for ShangRing procedure among study MC providers | An expected average of six months after study initiation
  Providers will complete a second questionnaire at the end of the study after all follow-up visits are completed. Study circumcision providers will be interviewed using a standardized questionnaire that includes items on preference for ShangRing.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Feldblum, Ph.D., Principal Investigator — FHI 360
Locations (2):
- Malawi (2):
  - Christian Health Association of Malawi, Lilongwe
  - St Gabriel's Hospital, Namitete